CLINICAL TRIAL: NCT03746093
Title: Effects of Non-alcoholic Beer in Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Effects of Non-alcoholic Beer in Patients With Type 2 Diabetes
Acronym: DIABEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIABEER
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants will consume a bottle of water (330 ml) every day for 12 weeks.
  Interventions: Dietary Supplement: Water
- Non-alcoholic beer (Experimental): Participants will consume non-alcoholic beer (330 ml) every day for 12 weeks.
  Interventions: Dietary Supplement: Non-alcoholic beer

INTERVENTIONS:
Dietary Supplement: Water — Participants will consume a bottle of water (330 ml) every day for 12 weeks.
  Arms: Control Group
Dietary Supplement: Non-alcoholic beer — Participants will consume non-alcoholic beer (330 ml) every day for 12 weeks.
  Arms: Non-alcoholic beer

SUMMARY:
The aim of the study is to investigate the effects of non-alcoholic beer in patients with type 2 diabetes. Subjects will be divided into two groups: the control group, where participants will be consuming a bottle of water (330ml) every day for 12 weeks, and the intervention group, where participants will be consuming a bottle of non-alcoholic beer (330ml) for the same period.

DETAILED DESCRIPTION:
This is a parallel, controlled randomized trial. The study will compare the effect of non-alcoholic beer consumption with water, in patients with type 2 diabetes.

All patients from both groups will receive a personalized nutritional intervention and will be followed throughout the study by a certified nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with type 2 diabetes mellitus, according to the American Diabetes Association criteria;
* Ages 40-80 years;
* Non-smoker;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Changes in oral glycaemic-control medications in the last 3 months;
* Subjects with HbA1c levels under 6.4% or above 10%;
* Subjects under insulinotherapy;
* Subjects with triglycerides levels above 4.52 nmol/L(400 mg/dL);
* Intake of antibiotics in the last 12 weeks;
* Subjects not willing to avoid drinking beer during the study;
* Subjects with a diagnosis of any digestive disease including functional bowel disorders such as IBS;
* Pregnant women or women planning to become pregnant during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in fasting capillary blood glucose from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in fasting insulin levels from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in HOMA-IR from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in HOMA-B from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in HbA1c levels from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)

SECONDARY OUTCOMES:
Changes in intestinal microbiota from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
  Bacterial DNA will be extracted from fecal samples. 16SRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Changes in body mass index from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
  Weight and height will be combined to report BMI in kg/m^2
Changes in total body fat mass from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in fasting serum total cholesterol from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in fasting serum high-density lipoprotein (HDL) cholesterol from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in fasting serum low-density lipoprotein (LDL) cholesterol from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)
Changes in fasting serum triglycerides from baseline to visit 2 and 3 | at visit 1 (after 1-week run-in period), visit 2 (after 6-week intake period), visit 3 (after 12-week intake period)

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School, NOVA University of Lisbon, Lisbon, Portugal